CLINICAL TRIAL: NCT01452581
Title: Liberal Versus Restrictive Transfusion During Symptomatic Moderate Anemia After Hip Arthroplasty
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of enrollment
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Oeivind Jans, M.D, Clinical Assitant, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: H-4-2011-058
Record Dates: First submitted 2011-10-10; First posted 2011-10-17 (Estimated); Last update posted 2015-03-06 (Estimated); Status verified 2015-03

CONDITIONS: Arthroplasty, Hip
Keywords: Transfusion; Red blood cells; Postoperative; Dizziness; Hip Arthroplasty
MeSH Terms: conditions — Dizziness | interventions — Erythrocyte Transfusion; HES 130-0.4

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- RBC transfusion (Active Comparator): Administration of up to 2 RBC units on the first postoperative day.
  (1 unit at a time followed by evaluation of the primary outcome measure)
  Interventions: Other: Red blood cell transfusion
- Restrictive: Colloid infusion (Placebo Comparator): Infusion of up to 2 x 280 ml colloid (6% Hydroxyethyl Starch 130/0.4 in 0.9% Sodium Chloride). 280 ml at a time. Evaluation of primary outcome after each intervention.
  Interventions: Drug: Voluven

INTERVENTIONS:
Other: Red blood cell transfusion — Maximal 2 units of packed red blood cells given one at a time on the first postoperative day. Evaluation of primary outcome is done after administration of each unit.
  Arms: RBC transfusion
Drug: Voluven — Infusion of up to 2 x 280 ml colloid (6% Hydroxyethyl Starch 130/0.4 in 0.9% Sodium Chloride). 280 ml at a time. Evaluation of primary outcome after each intervention.
  Arms: Restrictive: Colloid infusion

SUMMARY:
The purpose of this study is to evaluate the effects of transfusion of red blood cells in treating postoperative dizziness in patients with moderate postoperative anemia after total hip arthroplasty.

DETAILED DESCRIPTION:
Hip arthroplasty is associated with bleeding and postoperative anemia. However, the optimal strategy for transfusing red blood cells (RBC) remains to be elucidated. Postoperative anemia may cause dizziness and fatigue which delays early mobilization after surgery and may trigger the transfusion of one or more RBC units. However, it is not known whether the administration of 1-2 units of RBC to patients suffering from moderate postoperative anemia (HB 7.5 - 10 g/dl) will improve postoperative dizziness.

Thus, this randomized controlled study aims to evaluate whether the administration of 1-2 RBC units on the first postoperative day improves postoperative dizziness in patients undergoing total hip arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 and able to give consent
* Hip arthroplasty or hip revision arthroplasty
* Haemoglobin > 4.8 mmol/L and < 6.0 mmol/L on the first postoperative day
* Dizziness score ≥ 2.

Exclusion Criteria:

* Large ongoing bleeding
* Has already received RBC during the current admission
* New onset of cardiac arrhythmia suspected to be related to anemia
* Severe ischemic heart disease
* Renal failure with dialyses or oligouria / anuria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2011-10; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Postoperative Dizziness scale | Day 1 after surgery
  Dizziness scale (0-3) evaluated by the study nurse. The scale is evaluated upon information on the 1) severeness of dizziness AND 2) it´s consequenses for early mobilization after surgery.
  0 - No dizziness.
  1. - Light dizziness / No consequences for mobilization
  2. - Moderate dizziness / Only shorter periods of mobilization possible
  3. - Severe dizziness / No or only short bedside mobilization possible

SECONDARY OUTCOMES:
Timed up and go test (TUG) | Day 1 after surgery and on the day of discharge (expected mean 4 days after surgery)
  Measures the time it take the subject to rise from a chair, walk 3 meters and return to the chair.
Fatigue score | Day 1 after surgery and on the day of discharge (expected mean 4 days after surgery)
  Numeric rating scale 0-10, measuring subjective feeling of fatigue.
FACT-Anemia scale | 7 and 14 days
  Validated subjective score addressing anemia related symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Oeivind Jans, MD, Principal Investigator — Rigshospitalet, Denmark
Locations (2):
- Denmark (2):
  - Gentofte Hospital, Department of orthopedic surgery, Gentofte Municipality
  - Vejle Sygehus, Department of orthopedic surgery, Vejle